CLINICAL TRIAL: NCT02560597
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Epilepsy - Case Study in Patients With Epilepsia Partialis Continua (EPC) and Refractory Status Epilepticus (SE)
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Epilepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitement and finalisation of research on this topic by investigator
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kristl Vonck, Prof. Dr. Boon, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC2015/0083
Record Dates: First submitted 2015-09-18; First posted 2015-09-25 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Epilepsia Partialis Continua; Status Epilepticus
Keywords: epilepsy; epilepsia partialis continua; status epilepticus; treatment resistant; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Epilepsia Partialis Continua; Status Epilepticus; Epilepsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- repetitive transcranial magnetic stimulation (Experimental): rTMS delivered over the epileptogenic focus
  Interventions: Procedure: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation — Stimulation over the epileptogenic focus using variable stimulation protocols as described in literature. This protocol may vary case by case, depending on patient characteristics and achieved effect from previous stimulation.
  In absence of effect, rTMS is given on 5 consecutive days at most.

SUMMARY:
The purpose of this study is to assess the effects of repetitive transcranial magnetic stimulation (rTMS) as a treatment for Epilepsia Partialis Continua (EPC) or refractory Status Epilepticus (SE), when standard clinical treatments have failed.

DETAILED DESCRIPTION:
1. Study design:

   This is a case study, including up to 10 patients with EPC or refractory SE that are admitted to the service in the coming 5 years.

   If circumstances permit so, a baseline evaluation of seizure frequency over 1 week and a 24-hour baseline EEG registration will be obtained, as well as a baseline clinical neurologic exam. In case of therapeutic urgency, these baseline measurements will be omitted.

   The treatment itself consists of multiple stimulation sessions over multiple days, decided upon based on patient characteristics and the obtained effects. In absence of the desired effect, treatment will be repeated during 5 consecutive days at most.

   Patients will be followed-up clinically and electrographically. In case of therapeutic success, the treatment can be repeated over time when seizures reoccur.
2. Objectives:

   The primary objective of this study is to evaluate the effect of rTMS on the clinical status of patients with continuous refractory focal seizures (either EPC or SE). A beneficial effect on clinical status is defined as a decrease in seizure frequency or an interruption of continuous electrographic epileptiform activity, as well as an improvement in consciousness or other cortical functions that are disturbed by the EPC or SE (motor function, speech,...).

   As a secondary objective, the duration of the induced therapeutic effect will be evaluated, as well as the effect of rTMS on epileptiform discharges and the associated side effects and tolerability of the treatment.
3. Stimulation:

   The exact stimulation protocol will be decided upon case per case, based on similar reports in literature. The optimal stimulation protocol is currently unknown.
4. Rationale:

Patients with EPC often have a high number of debilitating seizures per day that are hard to control with anti-epileptic medication. Some cases of SE also do not respond to standard care and require heavy sedation of the patient.

Some of these patient may benefit from treatment with rTMS, which is painless, non-invasive and safe and can be administered at bedside. Moreover, in patients with EPC en SE, the (almost) continuous ictal activity allows an immediate effect evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsia partialis continua or refractory status epilepticus
* Prior investigations (EEG, MRI...) show a well-defined neocortical epileptogenic focus
* Informed consent signed by the patient or his/her legal representative

Exclusion Criteria:

* Pregnancy, short-term birth wish or childbearing age without adequate birth control
* Intracranial metal hardware (excluding dental filling): surgical clips, shrapnell, electrodes under the stimulation area
* Presence of pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants or deep brain stimulation (DBS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Seizure diary | Throughout the study, lasting approximately 4 weeks
  Self-reported seizure frequency throughout the study as a measure of clinical efficacy.
Electrographic epileptiform activity | Throughout the study, lasting approximately 4 weeks, with assessment before treatment (if possible) and after treatment
  Interictal or continuous epileptiform activity on EEG is assessed throughout the study as a measure of clinical efficacy.
Neurological examination | Throughout the study, lasting approximately 4 weeks
  Neurological examination assessing consciousness and other cortical functions that are potentially disturbed by the EPC or SE (eg. motor function, speech,...) is performed throughout the study as a measure of clinical efficacy.

SECONDARY OUTCOMES:
Duration of the clinical effect | Throughout the study, lasting approximately 4 weeks or as long as the outlasting effect lasts
  In case a beneficial clinical effect is obtained, an assessment of the duration of this effect will be performed.
Adverse events | Throughout the study, lasting approximately 4 weeks
  Assessment of the adverse events associated with rTMS in EPC/SE.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Meurs, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Belgium

REFERENCES:
- [Background] Rotenberg A, Bae EH, Takeoka M, Tormos JM, Schachter SC, Pascual-Leone A. Repetitive transcranial magnetic stimulation in the treatment of epilepsia partialis continua. Epilepsy Behav. 2009 Jan;14(1):253-7. doi: 10.1016/j.yebeh.2008.09.007. Epub 2008 Oct 30. PMID 18832045
- [Background] Morales OG, Henry ME, Nobler MS, Wassermann EM, Lisanby SH. Electroconvulsive therapy and repetitive transcranial magnetic stimulation in children and adolescents: a review and report of two cases of epilepsia partialis continua. Child Adolesc Psychiatr Clin N Am. 2005 Jan;14(1):193-210, viii-ix. doi: 10.1016/j.chc.2004.07.010. PMID 15564059
- [Background] Misawa S, Kuwabara S, Shibuya K, Mamada K, Hattori T. Low-frequency transcranial magnetic stimulation for epilepsia partialis continua due to cortical dysplasia. J Neurol Sci. 2005 Jul 15;234(1-2):37-9. doi: 10.1016/j.jns.2005.03.035. PMID 15946689
- [Background] Liu A, Pang T, Herman S, Pascual-Leone A, Rotenberg A. Transcranial magnetic stimulation for refractory focal status epilepticus in the intensive care unit. Seizure. 2013 Dec;22(10):893-6. doi: 10.1016/j.seizure.2013.06.014. Epub 2013 Jul 19. PMID 23876929
- [Background] Thordstein M, Constantinescu R. Possibly lifesaving, noninvasive, EEG-guided neuromodulation in anesthesia-refractory partial status epilepticus. Epilepsy Behav. 2012 Nov;25(3):468-72. doi: 10.1016/j.yebeh.2012.07.026. Epub 2012 Sep 12. PMID 22981238
- [Background] Graff-Guerrero A, Gonzales-Olvera J, Ruiz-Garcia M, Avila-Ordonez U, Vaugier V, Garcia-Reyna JC. rTMS reduces focal brain hyperperfusion in two patients with EPC. Acta Neurol Scand. 2004 Apr;109(4):290-6. doi: 10.1046/j.1600-0404.2003.00222.x. PMID 15016013
- [Background] VanHaerents S, Herman ST, Pang T, Pascual-Leone A, Shafi MM. Repetitive transcranial magnetic stimulation; A cost-effective and beneficial treatment option for refractory focal seizures. Clin Neurophysiol. 2015 Sep;126(9):1840-2. doi: 10.1016/j.clinph.2014.12.004. Epub 2014 Dec 15. No abstract available. PMID 25573025